CLINICAL TRIAL: NCT00323089
Title: Thoracoscopic Resection of Subcentimetre Lung Nodules After Localization Using Percutaneous Inserted Platinum Microcoil Under CT Guidance: a Pilot Study
Brief Title: Removal of Lung Nodules After Being Marked With a Microcoil
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Richard Finley, Principal Investigator, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H02-70562; 04-0048 (Other Grant/Funding Number: BC Lung Association); 20R42080 (Other Grant/Funding Number: BC Lung Association)
Record Dates: First submitted 2006-05-08; First posted 2006-05-09 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Lung Cancer
Keywords: microcoil; subcentimetre nodules
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: Preoperative CT-Guided Microcoil Localization (CTML) and Fluoroscopic-Guided Video-Assisted Thoracoscopic (VATS) Wedge Resection of Small Peripheral Pulmonary Nodules (SPPN)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surgical Arm (Experimental): Preoperative CT-Guided Microcoil Localization (CTML) and Fluoroscopic-Guided Video-Assisted Thoracoscopic (VATS) Wedge Resection of Small Peripheral Pulmonary Nodules (SPPN)
  Interventions: Procedure: microcoil insertion and excision

INTERVENTIONS:
Procedure: microcoil insertion and excision — The objective of this study is to determine if subcentimetre pulmonary nodules can be accurately and safely excised by endoscopic stapling devices after they have been localized using CT and marked with a microcoil device.

SUMMARY:
The objective of this study is to determine if subcentimetre pulmonary nodules can be accurately and safely excised by endoscopic stapling devices after they have been localized using CT and marked with a microcoil device.

The addition of real-time CT imaging and insertion of platinum microcoil markers to the technique of video assisted thoracoscopic stapled resection of subcentimetre pulmonary nodules, will decrease the rate of open thoracotomies required to completely resect the nodules.

DETAILED DESCRIPTION:
Lung cancer is the most common cause of cancer death for both men and women in the industrialized world. Small cell lung cancer accounts for about 25% of lung cancers and is usually widespread when it first presents. The remaining 75% of lung cancers are collectively termed non-small cell lung cancers. When presentation is by symptoms or incidental discovery, about 50 to 60% of non-small cell lung cancers are parenchymal nodules or masses and 40 to 50% are bronchial or hilar. More than 50% of patients with non-small cell cancer will have distant metastases at the time of diagnosis and only 25% will be potentially resectable for cure.1 Overall survival at five years for lung cancer is approximately 15% and has not significantly improved over the last several decades. Prognosis for lung cancer is affected by many factors but one of the most important is the stage of the disease at presentation. Individuals with peripheral lesions less than 3 cm in diameter (T1) at presentation are ideal candidates for surgical resection and have the best outcomes, with 5-year survival rates as high as 60 to 80%.2 Patients with small subcentimeter pulmonary nodes may have even better survival with resection. Computed tomography can now detect cancers less than 4 mm in diameter, and it has been shown that resection of subcentimetre lung cancers results in a survival rate of up to 85%.3 However, Suzuki et al found 54% of 92 patients undergoing video assisted thoracoscopic excision of subcentimetre nodules, required conversion to a thoracotomy. Forty percent of those nodules were found to be malignant.4 The most common reason for this conversion was failure to localize the nodule using thoracoscopic visualization or palpation. Furthermore, univariate and multivariate analysis of eleven variables revealed that if the distance from the pleural surface was greater than 5 mm, the probability of failure to detect the nodule was 63%.

ELIGIBILITY:
Inclusion Criteria:

* subcentimetre lung nodule

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2003-04; Primary Completion 2017-12-30 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
pulmonary nodule excision with microcoil | 6 years
  Thoracotomy and excision rates

SECONDARY OUTCOMES:
Recurrence and death from lung cancer | 10 years
  Death or CT recurrence of lung cancer

CONTACTS AND LOCATIONS:
Overall Officials: Richard Finley, MD, Principal Investigator — The University of British Columbia
Locations (1):
- Richard Finley, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No